CLINICAL TRIAL: NCT00920920
Title: A International Study on MRI-guided Brachytherapy in Locally Advanced Cervical Cancer
Brief Title: An International Study on Magnetic Resonance Imaging (MRI)-Guided Brachytherapy in Locally Advanced Cervical Cancer
Acronym: EMBRACE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Aarhus University Hospital (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); KU Leuven (Other); Mount Vernon Hospital (Other); Institute of Oncology Ljubljana (Other); ARTI Institute for Radiation Oncology Arnhem (Unknown); Maastricht University Medical Center (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Tata Memorial Hospital (Other Government); Kaposvár University (Other); Medical College of Wisconsin (Other); Leeds Cancer Centre at St. James's University Hospital (Other); St. Olavs Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); British Columbia Cancer Agency (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); University of Alberta (Other); University of Iowa (Other); Kuopio University Hospital (Other); Oslo University Hospital (Other); Hospital of Navarra (Other)
Responsible Party: Principal Investigator, Richard Pötter, Principal investigator, Medical University of Vienna
Other Study IDs: EMBRACE 1
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer
Keywords: 3D-4D MRI-based Brachytherapy; Cervical Cancer; Multicenter Clinical Study; Locally advanced cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: 3D MRI-guided Brachytherapy — MRI-based 3D-4D brachytherapy in locally advanced cervical cancer

SUMMARY:
Background:

The standard treatment of locally advanced cervical cancer is radio-chemotherapy including external beam radiotherapy (EBRT), brachytherapy (BT) and concomitant chemotherapy with weekly Cisplatin. While image based conformal EBRT is routinely used, prescription and reporting of BT is still based on specific dose points defined in 2D. Thus, for several decades the BT dose has most often been prescribed and reported to the Manchester point A defined according to different traditions.

Recently, a working group from GEC-ESTRO has published recommendations on contouring of tumour target and organs at risk (OAR) as well as on dose volume parameters to be reported for image guided BT in definitive radiotherapy for locally advanced cervical cancer. These recommendations are mainly derived from retrospective single institution experience with MRI based intracavitary BT. The major advantage of this technique is the possibility to conform the dose given by BT with regard to both volume (3D) and time (4D). Thus, by repetitive imaging performed before each BT implant it is possible adapt the dose given by BT to the anatomy of each individual patient taking into account not only the position of OAR but also the tumour regression which often is obtained by preceding EBRT and chemotherapy. Based on the experience collected so far, the image based BT approach is expected to have a major impact on the clinical outcome with a concomitant decrease in the rates of both local failure and morbidity.

Aims:

* To introduce MRI based 3D-4D BT in locally advanced cervical cancer in a multicenter setting within the frame of a prospective observational study.
* To establish a bench-mark for clinical outcome with image based BT in a large patient population with respect to local control, survival, morbidity and QoL
* To establish a reference material with regard to image based DVH parameters according to the guidelines from the GEC ESTRO working group.
* To correlate image based DVH parameters for CTV and for OAR with outcome
* To develop prognostic and predictive statistical models for clinical outcome including volumetric, dosimetric, clinical and biological risk factors
* To establish radiobiological parameter estimates that will allow a precise risk estimation in individual patients and aid in the development of new treatment protocols

DETAILED DESCRIPTION:
A prospective observational multicenter study will be performed in patients with locally advanced cervical cancer considered to be potentially curable by definitive radio-(chemo) therapy. The patients will be divided and analyzed in three strata according to risk of recurrence:

1. Small tumours
2. Large tumours favourable response
3. Large tumours with unfavourable response to the initial radio-(chemo) therapy.

A clinical local failure has to be validated by MRI and topographically correlated to the MRI based BT targets (HR CTV and IR-CTV) and the dose volume parameters of the treatment plan. It has to be classified as "inside", "at the edge", "outside".

Major events with regard to morbidity have to be reported using 3D imaging information integrating e.g. clinical examination, endoscopy and MRI. The location of organ damage (i.e. fistula) has to be identified in 3D and a correlation to the dose volume parameters for the affected region should be investigated.

Specific Aims

* To assess prospectively outcome for disease (local control, survival), for morbidity and for QoL life applying appropriate clinical, imaging and QoL protocols.
* To test that there are three groups representing different risks of recurrence: small tumours; large tumours with favourable response; large tumours with unfavourable response to initial radio-(chemo)therapy.
* To correlate local control (survival) and dose volume parameters for GTV and CTV for the overall cohort and for the 3 different risk groups and to establish hazard ratios and dose effect curves for the primary tumour.
* To correlate outcome data and dose volume parameters for the different OAR (rectum, sigmoid, bladder) and to establish hazard ratios and dose effect curves for OAR.
* To correlate QoL outcome to morbidity outcome.
* To quantify the change in DVH parameters obtained by image guided dose optimization of BT in the individual patient.
* To compare volumetric data on GTV and CTV at diagnosis and during treatment and relate them to dose volume parameters within the 3 different risk groups of the overall patient cohort.
* To evaluate the indicators for quality assessment throughout the whole study period in order to define systematic and random variations for the different indicators (e.g. contouring, applicator reconstruction, dose volume assessment).
* To validate from clinical outcome data the radiobiological equivalence calculations used for assessing dose and volume parameters in gynaecological radiotherapy.
* To test if the GYN GEC ESTRO recommendations for BT in cervical cancer are feasible in a multi-centre setting.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the uterine cervix considered suitable for curative treatment with definitive radio-(chemo)therapy including MRI guided BT
* Positive biopsy showing squamous-cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix.
* Staging according to FIGO and TNM guidelines
* MRI of pelvis at diagnosis is performed
* MRI, CT or PET-CT of the retroperitoneal space and abdomen at diagnosis is performed
* MRI with the applicator in place at the time of (first) BT will be performed
* Para-aortic metastatic nodes below L1-L2 are allowed
* Patient informed consent

Exclusion Criteria:

* Other primary malignancies except carcinoma in situ of the cervix and basal cell carcinoma of the skin
* Metastatic disease beyond para-aortic region (L1-L2)
* Previous pelvic or abdominal radiotherapy
* Previous total or partial hysterectomy
* Combination of preoperative radiotherapy with surgery
* Patients receiving BT only
* Patients receiving EBRT only
* Patients receiving neoadjuvant chemotherapy
* Contra indications to MRI
* Contra indications to BT
* Active infection or severe medical condition endangering treatment delivery
* Pregnant, lactating or childbearing potential without adequate contraception

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients to be included:
  Patients with newly biopsy proven squamous carcinoma, adenocarcinoma or adeno-squamous carcinoma of the uterine cervix, FIGO stage IB, IIA, IIB, IIIA, IIIB and IVA in whom definitive radiotherapy with curative intent is planned are qualified for the study. Patients with para-aortic metastatic nodes (stage IVB) to the level of L2 are also eligible but patients with further dissemination are not.
  Staging should as a minimal include gynaecological examination, MRI of the pelvis, abdominal CT or MRI and chest radiography. Further investigations are applied if necessary (e.g. cystoscopy, rectoscopy) or normally done according to institutional practice (e.g. PET-CT).
Sampling Method: Probability Sample
Enrollment: 1416 (Actual)
Dates: Start 2008-07; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
local control/morbidity | 5 years

SECONDARY OUTCOMES:
regional control | 5 years
disease free survival | 5 years
overall survival | 5 years
quality of life (QoL) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pötter, Prof., M.D., Principal Investigator — Department of Radiotherapy, Medical University of Vienna
Locations (1):
- MUV, Vienna, Austria

REFERENCES:
- [Derived] Schmid MP, Lindegaard JC, Mahantshetty U, Tanderup K, Jurgenliemk-Schulz I, Haie-Meder C, Fokdal LU, Sturdza A, Hoskin P, Segedin B, Bruheim K, Huang F, Rai B, Cooper R, van der Steen-Banasik E, Van Limbergen E, Pieters BR, Petric P, Ramazanova D, Ristl R, Kannan S, Hawaldar R, Ecker S, Kirchheiner K, Tan LT, Nout R, Nesvacil N, de Leeuw A, Potter R, Kirisits C; EMBRACE Collaborative Group. Risk Factors for Local Failure Following Chemoradiation and Magnetic Resonance Image-Guided Brachytherapy in Locally Advanced Cervical Cancer: Results From the EMBRACE-I Study. J Clin Oncol. 2023 Apr 1;41(10):1933-1942. doi: 10.1200/JCO.22.01096. Epub 2023 Jan 4. PMID 36599120
- [Derived] Potter R, Tanderup K, Schmid MP, Jurgenliemk-Schulz I, Haie-Meder C, Fokdal LU, Sturdza AE, Hoskin P, Mahantshetty U, Segedin B, Bruheim K, Huang F, Rai B, Cooper R, van der Steen-Banasik E, Van Limbergen E, Pieters BR, Tan LT, Nout RA, De Leeuw AAC, Ristl R, Petric P, Nesvacil N, Kirchheiner K, Kirisits C, Lindegaard JC; EMBRACE Collaborative Group. MRI-guided adaptive brachytherapy in locally advanced cervical cancer (EMBRACE-I): a multicentre prospective cohort study. Lancet Oncol. 2021 Apr;22(4):538-547. doi: 10.1016/S1470-2045(20)30753-1. PMID 33794207
- See also: Official homepage of the EMBRACE study — http://www.embracestudy.dk